CLINICAL TRIAL: NCT00253851
Title: Multi-centre, Double-blind, Randomized, Controlled Trial Comparing Intra-operative Regional Heparinization to Placebo for the Prevention of Deep Vein Thrombosis Following Total Knee Arthroplasty
Brief Title: Does Thinning the Blood During Surgery Prevent Blood Clots Following Total Knee Replacement Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: OHREB 2002597-01H
Record Dates: First submitted 2005-11-10; First posted 2005-11-15 (Estimated); Last update posted 2012-04-17 (Estimated); Status verified 2012-04

CONDITIONS: DVT; Osteoarthritis
Keywords: DVT; Osteoarthritis; Total Knee Arthroplasty
MeSH Terms: conditions — Osteoarthritis | interventions — Heparin

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: unfractionated heparin — Five minutes prior to tourniquet inflation, patients will receive 0.1 ml/kg/minute of intravenous (IV) unfractionated heparin (1000 units/ml) or placebo (normal saline solution). Five minutes will be allowed to elapse to ensure complete systemic heparinization. The operated limb will then be elevated and exsanguinated using an Esmarch bandage. Following cuff inflation, the contents of a second syringe will be administered IV over a 5 minute period. The second syringe will contain either protamine sulfate (1.0 mg/kg) to reverse the systemic heparin for patients in the treatment group, or normal saline for the control group. Study drugs will be administered by the anaesthesiologist via a peripheral IV. This new method of intraoperative regional heparinization has been used in two previous studies (Giachino et al., 2001; Giachino et al., 1985) with no adverse effects noted.

SUMMARY:
The goal of this study is to prevent blood clots from forming during surgery and a few days after total knee replacement surgery. This study will help us identify whether using a blood thinner in the operating room will stop blood clots from forming during the operation.

DETAILED DESCRIPTION:
Venous thromboembolism is a major cause of morbidity and mortality after lower limb orthopaedic surgery in the adult patient. If, as suggested, DVT formation begins intra-operatively then targeting this period to prevent clot formation could substantially reduce DVT rates in the TKA population. The present study aims to determine whether this intra-operative regional heparinization technique is effective in preventing the intra-operative formation of DVT following TKA, as evidenced by venography in the early post-operative period.

ELIGIBILITY:
Inclusion Criteria:

1. Undergoing unilateral primary total knee arthroplasty
2. Males and non-pregnant females ages 18-90 (pre-menopausal females will undergo a serum pregnancy test at screening)
3. Full weight bearing status (of non-operated leg) following surgery
4. Patient able to understand and willing to sign informed consent

Exclusion Criteria:

* 1) Known hypersensitivity to contrast media 2) Patients taking Metformin 3) Serum creatinine above 180Fmol/L 4) Platelets < 100 x 10 9/L, INR/PTT > 1.5 x normal 5) History of heparin induced thrombocytopenia 6) Allergy to heparin or fish 7) Prior use of protamine sulfate (i.e., protamine-containing insulin) 8) Vasectomized or infertile males 9) History of bleeding disorder 10) Bilateral total knee arthroplasty 11) History of stroke or myocardial infarction in previous 6 months 12) Traumatic spinal anaesthesia (two or more attempts and/or bloody) 13) History of previous DVT/PE 14) Active peptic ulcer disease (e.g., GI bleed, rectal bleed) 15) Currently on chronic anticoagulant therapy 16) Contra-indication to heparin 17) Patient is taking part in any other investigational study 18) Previous contralateral TKR or hip replacement

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2003-07; Primary Completion 2011-05 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
DVT as determined by venography | 5 day post op

SECONDARY OUTCOMES:
Bleeding rate Rate of PE Complication Rate | 2 week post op

CONTACTS AND LOCATIONS:
Overall Officials: A Giachino, Principal Investigator — OHRI
Locations (1):
- Ottawa Hospital, Ottawa, Ontario, Canada